CLINICAL TRIAL: NCT06494930
Title: The Effect of Functional Respiratory Muscle Training on Respiratory Function and Physical Performance in Football Players
Brief Title: The Effect of Functional Respiratory Muscle Training on Respiratory Function and Physical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yunus Emre Tutuneken, PhD, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12
Record Dates: First submitted 2024-06-02; First posted 2024-07-10 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Muscle; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F-IMT Group (Experimental): Participants in this group will perform functional IMT under supervision 5 days a week. In functional IMT, the core stabilization exercise protocol will be applied at the same time as the participants practice the breathing exercise with the device.
  Interventions: Other: F-IMT
- Control Group (Active Comparator): Participants in this group will also apply a core stabilization exercise protocol under supervision 5 days a week.
  Interventions: Other: Core Stabilization Exercise

INTERVENTIONS:
Other: F-IMT — A core stabilization exercise protocol including functional respiratory muscle training will be applied to the F-IMT group. IMT will be provided with the red Powerbreath Plus MR exercise device. Initial training intensity will be set at 50% of the MIP value measured at the athlete's first evaluation. Every two weeks, the athlete will be re-evaluated the new MIP value will be measured, and the training intensity will be adjusted to 50% of the newly measured MIP value. After the nose clip is attached, the athlete will be asked to take the device's mouthpiece into his mouth, close his lips tightly, and take a deep, fast, and powerful breath, then exhale slowly and completely with minimal effort. While the athlete does breathing exercises with the device, he will also do core stabilization exercises. Athletes will be asked to train 30 minutes daily, five days a week, for six weeks.
  Arms: F-IMT Group
Other: Core Stabilization Exercise — Only the core stabilization exercise protocol will be applied to the control group. Athletes will be asked to train 30 minutes a day, five days a week, for six weeks.
  Arms: Control Group

SUMMARY:
The study aims to investigate the effects of core stabilization exercise, which includes functional respiratory muscle training, on respiratory function, aerobic capacity, trunk stabilization, and physical performance in football players.

Licensed athletes who actively engage in sports and play football will be included in the project. Volunteers included in the study will be randomly divided into two groups: study and control groups. Different methods will be used in the study for respiratory function testing, respiratory muscle strength measurement, trunk stabilization evaluation, and performance evaluation. To apply these methods, a spirometer device (according to ATS/ERS criteria with Cosmed Pony FX, Italy), portable, electronic oral pressure measurement device (with Micro Medical Micro RPM, Rochester, England), Plank and Sorenson tests will be used. A core stabilization exercise protocol including functional respiratory muscle training will be applied to the study group. The control group will only apply the same core stabilization exercise protocol as the study group.

This study aims to investigate the effects of functional respiratory muscle training and to add it to the training program of athletes according to the results.

DETAILED DESCRIPTION:
Football is a sport branch that requires a high degree of coordination, using motoric properties such as general endurance and coordination, as well as aerobic and anaerobic efforts. Studies argue that core strength positively affects athletic performance, reduces the risk of injury, and has an effect on the treatment of pain in the back area. Core stability is very important in terms of sports performance. Respiratory functions of all athletes, regardless of sports branches; It varies depending on physiological, functional, and psychological factors. Because disruption of respiratory muscle functions or respiratory muscle fatigue is a factor that jeopardizes the exercise performance of athletes. Numerous studies have shown that respiratory muscle training reduces respiratory muscle fatigue and sympatho-excitation during intense exercise. Previous studies focusing on the effects of respiratory muscle training have shown increased respiratory muscle strength in triathletes and marathon runners, rowers, cyclists, and divers. There are a limited number of studies investigating the effect of respiratory muscle training on football players. Our study, based on research in recent literature, aims to investigate the effects of core stabilization exercise, which includes functional respiratory muscle training, on respiratory function, aerobic capacity, trunk stabilization, and physical performance in football players.

Licensed athletes who actively engage in sports and play football will be included in the project. Volunteers included in the study will be randomly divided into two groups: study and control groups. Different methods will be used in the study for respiratory function test (PFT), measurement of respiratory muscle strength, trunk stabilization evaluation, and performance evaluation. To apply these methods, a spirometer device (according to ATS/ERS criteria with Cosmed Pony FX, Italy), portable, electronic oral pressure measurement device (with Micro Medical Micro RPM, Rochester, England), Plank and Sorenson tests will be used. A core stabilization exercise protocol including functional respiratory muscle training will be applied to the study group. The control group will only apply the same core stabilization exercise protocol as the study group.

This study aims to investigate the effects of functional respiratory muscle training and to add it to the training program of athletes according to the results. Aiming to improve the health and working dynamics of the respiratory muscles in athletes by applying functional muscle training to participants, as well as showing its effect on instant and prospective performance in athletes, is the ultimate goal to be shaped by the study findings. The study will shed light on this aspect with its functioning and method for researchers in the field. With the analysis and presentation of the data obtained from our study, the gaps in the current literature will be filled.

ELIGIBILITY:
Inclusion Criteria:

Professional or recreational athlete Must be approved participation Must be ability to cooperate with the exercise training and evaluation methods to be applied

Exclusion Criteria:

Have surgery within the last six months Cardiovascular or pulmonary disease Taking a break from sports

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
İnspiratory muscle strength measurement | 6 week
  The athletes' maximum inspiratory intraoral pressure (MIP) will be measured by a portable, electronic oral pressure measuring device, and the values will be recorded in cmH2O.
Plank Test | 6 week
  Subjects are asked to lie face down, stand on their toes with their forearms and elbows bilaterally shoulder-width apart, lift the pelvis, and form a straight line parallel to the floor with their neck, shoulders, back, hips, and legs, and the subject maintains this posture. Once the time starts, the time until the subject gets tired and/or breaks his posture is recorded in seconds.
Sorenson Test | 6 week
  For this test, the athlete will be laid face down with his body hanging off the bed from the anterior superior iliac spine. The athlete is asked to keep his body parallel to the ground against gravity, with his legs fixed at the gastrocnemius muscle level and his hands clasped on his chest. Partial trunk extension is allowed. When posture is impaired and/or the athlete quits the experiment due to fatigue and pain, the time is stopped and the score in seconds is recorded.
Y Balance Test | 6 week
  The "Y Balance Test" platform will be used to measure dynamic postural control. Each participant's leg length will be recorded in centimeters by measuring bilaterally in the supine position from the anterior superior iliac point to the distal part of the medial malleolus. Measurements will be tested barefoot, in 3 directions, with ANT reaching as the distance between the participant's central toe tip and PL and PM as the distance between the farthest point the participant can reach from the heel of the foot.
Ekspiratory muscle strength measurement | 6 week
  The athletes' maximum expiratory intraoral pressure (MEP) will be measured by a portable, electronic oral pressure measuring device, and the values will be recorded in cmH2O.

SECONDARY OUTCOMES:
The forced vital capacity (FVC) | 6 week
  In the respiratory function test, the athletes' forced vital capacity (FVC) will be measured with a portable spirometer. Pulmonary function test parameters will be expressed in liters and percentage of the expected value. Respiratory function test will be performed with a spirometer device according to ATS/ERS criteria.
The forced expiratory volume in the first second (FEV1) | 6 week
  In the respiratory function test, the athletes' forced expiratory volume in the first second (FEV1) will be measured with a portable spirometer. Pulmonary function test parameters will be expressed in liters and percentage of the expected value. Respiratory function test will be performed with a spirometer device according to ATS/ERS criteria.
The forced expiratory volume in the first second to forced vital capacity (FEV1/FVC) | 6 week
  In the respiratory function test, the athletes' ratio of forced expiratory volume in the first second to forced vital capacity (FEV1/FVC) will be measured with a portable spirometer. Pulmonary function test parameters will be expressed in liters and percentage of the expected value. Respiratory function test will be performed with a spirometer device according to ATS/ERS criteria.
The peak flow rate (PEF) | 6 week
  In the respiratory function test, the athletes' peak flow rate (PEF) will be measured with a portable spirometer. Pulmonary function test parameters will be expressed in liters and percentage of the expected value. Respiratory function test will be performed with a spirometer device according to ATS/ERS criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Yunus Emre TÜTÜNEKEN, Istanbul, Zeytinburnu, Turkey (Türkiye)